CLINICAL TRIAL: NCT05859698
Title: A Phase 4, Single-Arm, Open-Label Study to Evaluate the Effectiveness of Valbenazine on Patient- and Clinician-Reported Outcomes in Subjects With Tardive Dyskinesia
Brief Title: Study of the Effectiveness of Valbenazine on Patient- and Clinician-Reported Outcomes in Participants With Tardive Dyskinesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NBI-98854-TD4020
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Results first posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2025-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depressive Disorder; Tardive Dyskinesia
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major; Tardive Dyskinesia | interventions — valbenazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Valbenazine (Experimental): Valbenazine administered once daily for 24 weeks.
  Interventions: Drug: Valbenazine

INTERVENTIONS:
Drug: Valbenazine — Valbenazine capsules for oral administration
  Other Names: NBI-98854

SUMMARY:
This study will evaluate the effectiveness of valbenazine on patient- and clinician-reported outcomes assessing health-related quality of life, functioning, and treatment effect in participants with tardive dyskinesia (TD) who are receiving valbenazine for up to 24 weeks.

ELIGIBILITY:
Key Inclusion Criteria:

* At least 18 years of age
* Have one of the following clinical diagnoses: schizophrenia or schizoaffective disorder, bipolar disorder, or major depressive disorder
* Have a clinical diagnosis of neuroleptic-induced TD
* Medication(s) for schizophrenia or schizoaffective disorder, bipolar disorder, or major depressive disorder and other protocol-allowed concurrent medications must be at a stable dose and expected to remain stable during the study
* Participants must be outpatients and have a stable psychiatric status

Key Exclusion Criteria:

* Have comorbid abnormal involuntary movement(s) (for example, Parkinsonism, akathisia) that is more prominent than TD
* Have an active, clinically significant unstable medical condition in the judgement of the investigator, or have any laboratory value outside the normal range that is considered by the investigator to be clinically significant at the screening visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-12-27 (Actual); Study Completion 2024-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Lead, Study Director — Neurocrine Biosciences
Locations (18):
- United States (18):
  - Neurocrine Clinical Site, Bryant, Arkansas
  - Neurocrine Clinical Site, Anaheim, California
  - Neurocrine Clinical Site, Orange, California
  - Neurocrine Clinical Site, Torrance, California
  - Neurocrine Clinical Site, Bonita Springs, Florida
  - Neurocrine Clinical Site, Miami, Florida
  - Neurocrine Clinical Site, Miami Lakes, Florida
  - Neurocrine Clinical Site, Okeechobee, Florida
  - Neurocrine Clinical Site, Tampa, Florida
  - Neurocrine Clinical Site, Atlanta, Georgia
  - Neurocrine Clinical Site, Augusta, Georgia
  - Neurocrine Clinical Site, Marietta, Georgia
  - Neurocrine Clinical Site, Lincoln, Nebraska
  - Neurocrine Clinical Site, Beechwood, Ohio
  - Neurocrine Clinical Site, Oklahoma City, Oklahoma
  - Neurocrine Clinical Site, DeSoto, Texas
  - Neurocrine Clinical Site, El Paso, Texas
  - Neurocrine Clinical Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results are reported for the overall population as a single arm irrespective of dose, as pre-specified in the protocol. Individual participants could receive different dose levels over the duration of the treatment period.
Groups:
- Valbenazine: Participants received valbenazine oral capsules once a day (qd) at a dose of either 40 milligrams (mg), 60 mg or 80 mg for up to 24 weeks.
Period: Overall Study
Arm/Group | Valbenazine
Started | 59
Received at Least 1 Dose of Valbenazine | 59
Completed | 51
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 2
Not completed — Other Than Specified | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Valbenazine: Participants received valbenazine oral capsules qd at a dose of either 40 mg, 60 mg or 80 mg for up to 24 weeks.
Arm/Group | Valbenazine
Number analyzed (Participants) | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (11.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24
  Not Hispanic or Latino | 35
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Black or African American | 17
  White | 38
  Native Hawaiian or Other Pacific Islander | 0
  Other | 2
  Multiple | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Tardive Dyskinesia Impact Scale (TDIS) Total Score at Week 24
Description: The TDIS assesses the impact of impairment and disability associated with dyskinesia. It defines impact of tardive dyskinesia (TD) in terms of 6 scales: Mouth/Throat Function (3 items), Dexterity (2 items), Mobility (2 items), Pain (1 item), Emotional (2 items), and Social (1 item). Each item measured the impact of dyskinetic movements in terms of difficulty or frequency over the last 7 days on a 5-point scale, with scores ranging from 0 to 4. Response options for the difficulty items ranged from not at all (0) to extremely (4); those for the frequency items ranged from never (0) to all of the time (4). The TDIS total score was the sum of the scores of TDIS Items 1 to 11. Total scores ranged from 0 to 44, with higher scores representing greater TD impact.
Time Frame: Baseline, Week 24
Population: The Full Analysis Set included all enrolled participants with at least one baseline efficacy data point for any measure and at least one postbaseline efficacy data point for any measure. Here, "Overall Number of Participants Analyzed" = the number of participants evaluable at the timepoint assessed.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Valbenazine
Number analyzed (Participants) | 45
score on a scale | -8.0 [-10.48 to -5.44]

2. Primary Outcome: Change From Baseline in the Sheehan Disability Scale (SDS) Items 1, 2, and 3 Score at Week 24
Description: The SDS included 3 self-rated items designed to measure how work, social life, and family life are impaired by current psychiatric symptoms. Each item includes an 11-point analog scale that uses visual-spatial, numeric, and verbal descriptive anchors to represent the degree of disruption from 0 (none at all) to 10 (extremely). Participants who had not worked for pay or attended school in the previous 7 days for reasons unrelated to TD did not respond to Item 1 and were therefore excluded from the analysis of that item.
Time Frame: Baseline, Week 24
Population: The Full Analysis Set included all enrolled participants with at least one baseline efficacy data point for any measure and at least one postbaseline efficacy data point for any measure. Here, "Overall Number of Participants Analyzed" = the number of participants evaluable at the timepoint assessed. "Number Analyzed" = participants evaluable for specified SDS item.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Valbenazine
Number analyzed (Participants) | 45
score on a scale
  Item 1: Work/School Impairment: number analyzed (Participants) | 10
  Item 1: Work/School Impairment | -1.2 [-2.98 to 0.58]
  Item 2: Social Life Impairment | -2.3 [-3.23 to -1.43]
  Item 3: Family Life/Home Responsibilities | -1.6 [-2.54 to -0.57]

3. Primary Outcome: Change From Baseline in the Euro Quality of Life Visual Analogue Scale (EQ-VAS) Score at Week 24
Description: Participants rated their overall health on a 0 to 100 hash-marked, vertical EQ-VAS where 0 represents 'The worst health you can imagine' and 100 represents 'The best health you can imagine.' An increase from baseline indicates an increase in overall health.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Valbenazine
Number analyzed (Participants) | 45
score on a scale | 13.1 [7.70 to 18.48]

4. Secondary Outcome: Patient Global Impression of Change (PGI-C) Score at Week 24
Description: Participants rated the change in their TD symptoms from the initiation of study treatment dosing by choosing one of 7 responses (1=very much improved, 2=much improved, 3=minimally improved, 4=not changed, 5=minimally worse, 6=much worse, and 7=very much worse). Number of participants with PGI-C score responses are reported.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Valbenazine
Number analyzed (Participants) | 45
Participants
  1 = Very Much Improved | 13
  2 = Much Improved | 19
  3 = Minimally Improved | 10
  4 = Not Changed | 2
  5 = Minimal Worse | 1
  6 = Much Worse | 0
  7 = Very Much Worse | 0

5. Secondary Outcome: Change From Baseline in the Clinical Global Impression of Severity - Tardive Dyskinesia (CGI-TD-S) Score at Week 24
Description: The CGI-TD-S is based on a 7-point scale (range; 1=normal, not at all ill to 7=among the most extremely ill patients), was used to rate the overall global severity of TD.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Valbenazine
Number analyzed (Participants) | 45
score on a scale | -1.47 [-1.8 to -1.2]

6. Secondary Outcome: Change From Baseline in the Abnormal Involuntary Movement Scale (AIMS) Dyskinesia Total Score at Week 24
Description: The AIMS dyskinesia total score was defined as the sum of the scores of AIMS items 1 through 7. The scores for each item ranged from 0 (no dyskinesia) to 4 (severe dyskinesia). If any of the seven items had a missing value, the total score for that participant/visit was set equal to missing. The AIMS dyskinesia total score can therefore range from 0 to 28, with higher scores indicating greater severity.
Time Frame: Baseline, Week 24
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Valbenazine
Number analyzed (Participants) | 45
score on a scale | -6.8 [-7.75 to -5.81]

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Description: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Valbenazine
All-Cause Mortality (participants affected / at risk) | 1/59
Serious Adverse Events (participants affected / at risk) | 6/59
Other Adverse Events (participants affected / at risk) | 6/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine (N=59)
Peptic ulcer (Gastrointestinal disorders) | 1
Chest pain (General disorders) | 1
Medication error (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Suicidal ideation (Psychiatric disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valbenazine (N=59)
Nausea (Gastrointestinal disorders) | 3
Somnolence (Nervous system disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2024-01-29): https://cdn.clinicaltrials.gov/large-docs/98/NCT05859698/Prot_000.pdf
  • Statistical Analysis Plan (2025-01-10): https://cdn.clinicaltrials.gov/large-docs/98/NCT05859698/SAP_001.pdf